CLINICAL TRIAL: NCT00366743
Title: Analysis of Visual Outcomes, Contrast Sensitivity, Glare, Induction of High Order Aberrations and Wavefront Technology, Following LASIK Surgery
Brief Title: Evaluation of Visual Outcomes After Myopic LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-05-001
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2005-06

CONDITIONS: Myopia; Astigmatism; Myopic Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

INTERVENTIONS:
Procedure: Conventional LASIK
Procedure: Wavefront-guided LASIK

SUMMARY:
The aim of the study was to evaluate visual outcomes, contrast sensitivity, glare testing and high order aberrations induced by different laser technologies and to evaluate differences in aberrometer technology. We hypothesized that there will not be differences among conventional or wavefront guided treatments.

DETAILED DESCRIPTION:
The aim of the study was to evaluate and compare visual outcomes, contrast sensitivity, glare testing and induction of high order aberrations by different laser technologies and to evaluate differences in aberrometer technology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Candidates for bilateral LASIK
* Myopic range: 0.00 to -7.00 D
* Astigmatism: 0.00 to -5.00 D

Exclusion Criteria:

* Pupil size greater than 8mm diameter, infrared measurement
* thin corneas (preoperatively calculated minimal residual bed < 250 um)
* irregular astigmatism
* asymmetric astigmatism
* unstable refraction
* other criteria that preclude the patient to undergo LASIK

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2003-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Visual acuity
Contrast sensitivity
Induction of high order aberrations

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Medical University of South Carolina